CLINICAL TRIAL: NCT02669862
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of A-101 Solution in Subjects With Common Warts.
Brief Title: A Study of A-101 Solution in Subjects With Common Warts.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-WART-201
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Common Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- A-101 Solution 40 (Experimental): A-101 Solution 40% administered once per week
  Interventions: Drug: A-101 Solution 40
- A-101 Solution 45 (Experimental): A-101 Solution 45% administered once per week
  Interventions: Drug: A-101 Solution 45
- Vehicle Solution (Placebo Comparator): Vehicle Solution administered once per week
  Interventions: Drug: Vehicle Solution

INTERVENTIONS:
Drug: A-101 Solution 40
  Arms: A-101 Solution 40
Drug: A-101 Solution 45
  Arms: A-101 Solution 45
Drug: Vehicle Solution
  Arms: Vehicle Solution

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel-group study with 3 treatment groups.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, parallel-group study with 3 treatment groups. During Visit 1, the Investigator will identify 1 eligible common wart on the trunk or extremities on each subject. The wart will be treated up to a maximum of 8 times at 1 week intervals during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject has a clinical diagnosis of common warts
3. Subject has 1 appropriate Target Wart as defined below, on the trunk or extremities:

   * Have a longest axis that is 3mm to 10mm
   * Have a thickness ≤3mm
   * Be a discrete lesion
   * Be, when centered in the circular cutout of the provided template, the only common wart present
   * Not be periungual, subungual, genital or anal
   * Not be covered with hair which, in the Investigator's opinion, would interfere with the study medication treatments or the study evaluations Not be in an area that may be occluded (by clothing, footwear or within a skin fold).
4. The Target Wart has a Physician Wart Assessment (PWA) ≥2
5. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an approved effective method of birth control for the duration of the study
6. Subject is non-pregnant and non-lactating
7. Subject is in good general health and free of any known disease state or physical condition which, in the Investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
8. Subject is willing and able to follow all study instructions and to attend all study visits
9. Subject is able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

1. Subject has clinically atypical warts on the trunk or extremities
2. Subject is immune compromised (due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant status, etc.)
3. Subject has a history of Human Immunodeficiency Virus (HIV) infection
4. Subject has had any Human Papilloma Virus (HPV) vaccine within 1 year prior to enrollment
5. Subject has used any of the following intralesional therapies within the specified period prior to enrollment to the Target Wart:

   * Immunotherapy (Candida antigen, mumps antigen, Trichophyton antigen);
   * Anti-metabolite therapy (bleomycin, 5-fluorouracil)
6. Subject has used any of the following systemic therapies within the specified period prior to enrollment:

   * Immunomodulatory/immunosuppressant therapy (e.g., etanercept, alefacept, infliximab);
   * Glucocortico-steroids (inhaled and intra-nasal steroids are permitted);
7. Subject has used any of the following topical therapies within the specified period prior to enrollment on, or in a proximity to the Target Wart, which in the Investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations:

   - LASER (pulsed-dye laser), light (intense pulsed light, photo-dynamic therapy, other energy based therapy); Immuno-therapy ( imiquimod, squaric acid dibutyl ester, etc.); Anti-metabolite therapy (5-fluorouracil); Retinoids; Liquid nitrogen, electrodesiccation, curettage; Over-the-counter wart therapies
8. Subject has had any of the following within the specified period prior to enrollment on, or in a proximity to the target lesion, which in the Investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations:

   * A cutaneous malignancy;
   * A pre-malignancy (actinic keratosis)
9. Subject has a history of sensitivity to any of the ingredients in the study medications
10. Subject has any current skin disease (psoriasis, atopic dermatitis, eczema, sun damage, etc.), skin condition (sunburn, open wounds) or other disease or condition (uncontrolled diabetes) which, in the Investigator's opinion, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
11. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-12-21; Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Aclaris Therapeutics, Inc.
Locations (1):
- Aclaris Therapeutics, Inc., Wayne, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 Solution 40: A-101 Solution 40% administered once per week
  A-101 Solution 40
- A-101 Solution 45: A-101 Solution 45% administered once per week
  A-101 Solution 45
- Vehicle Solution: Vehicle Solution administered once per week
  Vehicle Solution
Period: Overall Study
Arm/Group | A-101 Solution 40 | A-101 Solution 45 | Vehicle Solution
Started | 33 | 34 | 31
Completed (Patients completing visit 10 according to protocol) | 31 | 29 | 26
Not Completed | 2 | 5 | 5
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — moved | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-101 Solution 40 | A-101 Solution 45 | Vehicle Solution | Total
Number analyzed (Participants) | 33 | 34 | 31 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (16.40) | 41.2 (14.11) | 39.5 (13.37) | 40.7 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 17 | 52
  Male | 19 | 13 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Percentages are based on the number of randomized subjects within each treatment group.
  Participants
    Hispanic or Latino | 3 | 6 | 2 | 11
    Not Hispanic or Latino | 27 | 28 | 26 | 81
    Unknown or Not Reported | 3 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 2 | 3 | 8
  White | 30 | 32 | 27 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 31 | 98

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Based on Mean Change in Physician Wart Assessment Over Time
Description: The primary effectiveness will consist of the mean change from Visit 2 to Visit 10 in Physician Wart Assessment (PWA) performed using Analysis of Covariance (ANCOVA) with Visit 2 PWA as the covariate. Physician Wart Analysis is a measurement scale from 0 to 3 that evaluates the wart with 0 being clear and 3 being clinically diagnosable wart that is raised, with an obviously rough surface.
Time Frame: 57 Days
Population: Number of participants analyzed is the number of participants completing the protocol through visit 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | A-101 Solution 40 | A-101 Solution 45 | Vehicle Solution
Number analyzed (Participants) | 32 | 31 | 27
units on a scale | -0.38 (0.75) | -1.00 (0.97) | -0.44 (0.85)
Statistical Analysis 1: Comparison: A-101 Solution 40 vs Vehicle Solution; In this table Study Day 01 / Visit 2 has been considered as Baseline visit for calculating mean and mean change. PVal*- ANCOVA used for calculating P-value by comparing Vehicle against each Active treatment group using baseline values as the covariate; Test type: Other; p = 0.555, ANCOVA; Baseline values were the covariate
Statistical Analysis 2: Comparison: A-101 Solution 45 vs Vehicle Solution; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.009, ANCOVA — PVal*- ANCOVA used for calculating P-value by comparing Vehicle against each Active treatment group using baseline values as the covariate. No adjustments for multiple comparisons

2. Secondary Outcome: Durability of Response - Percentage of Participants That Were Clear at Visit 10 That Are Still Clear at Visit 13
Description: Percentage of subjects whose target wart was clear at Visit 10 and who remained clear at Visit 13 for active treatment groups
Time Frame: visit 10 to visit 13
Population: Only the number of participants clear at visit 10 are compared to the number of participants clear at visit 13 to get the percentage clear for active treatment groups only.
Measure: Number (95% Confidence Interval); unit: percentage participants
Arm/Group | A-101 Solution 40 | A-101 Solution 45
Number analyzed (Participants) | 1 | 8
percentage participants | 100 | 87.50 [64.58 to 99.99]

3. Secondary Outcome: PWA Responder
Description: The percentage of participants who were responders with the target wart judged to be clear (PWA = 0) at Visit 10.
Time Frame: Day 57
Population: PP population = participants completing protocol to visit 10
Measure: Number; unit: percentage of responders
Arm/Group | A-101 Solution 40 | A-101 Solution 45 | Vehicle Solution
Number analyzed (Participants) | 32 | 31 | 27
percentage of responders | 3.13 | 25.81 | 3.70
Statistical Analysis 1: Comparison: A-101 Solution 40 vs Vehicle Solution; PVal*- Chi-Square test used for calculating P-value by comparing Vehicle against each Active treatment group; Test type: Other; p = 0.9313, Chi-squared — Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: A-101 Solution 45 vs Vehicle Solution; Test type: Other; p = 0.0236, Chi-squared — Not adjusted for multiple comparisons

ADVERSE EVENTS:
Arm/Group | A-101 Solution 40 | A-101 Solution 45 | Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 8/33 | 6/34 | 10/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution 40 (N=33) | A-101 Solution 45 (N=34) | Vehicle Solution (N=31)
Application site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) — Administration site conditions
Seasonal allergy (Immune system disorders) | 1 (1) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of Sponsor.